CLINICAL TRIAL: NCT00647439
Title: Epigenetics, Molecular Genetics, and Biomarkers of Degenerative and Inflammatory Ocular Diseases
Brief Title: Genetics and Markers of Degenerative and Inflammatory Eye Diseases
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080099; 08-EI-0099
Record Dates: First submitted 2008-03-28; First posted 2008-03-31 (Estimated); Last update posted 2018-12-10 (Actual); Status verified 2018-12-04

CONDITIONS: Diabetic Retinopathy; Age-Related Macular Degeneration (AMD); Uveitis
Keywords: OCULAR INFLAMMATORY DISEASE; Immune Mediated; Gene Expression Patterns; Diabetic Retinopathy; Age-Related Macular Degeneration; AMD; Uveitis
MeSH Terms: conditions — Diabetic Retinopathy; Macular Degeneration; Uveitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
This study will identify genes that are associated with inflammation or degeneration of the retina (membrane lining the back of the eye that relays vision signals to the brain). It is thought that many retinal conditions are due to an altered immune system and are based on how the person s genes function and communicate.

People 4 years of age or older who have a retinal condition such as uveitis, age-related macular degeneration or diabetic retinopathy may be eligible for this study. Healthy volunteers and healthy people who have a family member with one of these conditions are also eligible. Patients with inherited retinal degeneration are excluded.

Participants undergo the following tests and procedures:

* Eye examination to assess visual acuity (eye chart test) and eye pressure, and to examine the pupils, lenses, retina and eye movements. Photographs of the inside of the eye may also be taken. The pupils are dilated with drops for this examination.
* Blood draw for genetic testing.

Participants may also undergo one or more of the following tests:

* Optical coherence tomography. This is a type of photograph of the back of the eye to measure thickness of the retina.
* Fluorescein angiography and indocyanine green angiography. Pictures of the eye s blood vessels are taken using either a fluorescein or indocyanine green dye. The dye is injected into a vein in an arm and travels to the blood vessels in the eyes. A camera takes pictures of the dye as it flows through the blood vessels.
* Electroretinogram (ERG) to measure retinal function. The patient sits in a dark room for 30 minutes with his or her eyes patched. Then, a small metal disk electrode is taped to the forehead, the eye patches are removed, the surface of the eye is numbed with eye drops, and contact lenses are placed on the eyes. The patient then watches flashing lights. The contact lenses sense small electrical signals generated by the retina when the light flashes....

DETAILED DESCRIPTION:
Objective:

This project will study epigenetic mechanisms, the inheritance of (both Mendelian and complex) and biomarkers of Immune Mediated Eye Diseases, in families of many nationalities and ethnic backgrounds in order to identify the genes that, when genetically mutated or epigenetically regulated, cause immune mediated eye disease, and the pathophysiology through which they act.

Study Population: The number of participants to be enrolled has no logical upper limit, but will be at 1,000 during the next five years. Race, age and sex matched controls, anonymous volunteers will also be needed to donate a blood sample. The study consists of ascertaining individuals and families with multiple individuals, if possible, affected by immune mediated ocular disease.

Design:

These patients and their families will undergo detailed ophthalmologic examinations and, where indicated, additional non-investigational examinations to characterize their ocular status. A blood sample will be collected from each individual and immunophenotyped using Flow Cytometry. Serum will be isolated for testing serological markers. One or more sub-populations of cells (including but not limited to CD4 plus and CD8 plus T cells, B cells, CD14 plus monocytes, dendritic cells, NK cells, neutrophils and granulocytes) will be isolated. DNA, RNA and chromatin may be isolated for further gene expression profiling and epigenetic studies. Association of genetic or epigenetic changes with ocular inflammatory disease in patients and their families will be identified using one of the techniques including but not limited to DNA-seq, BS-seq, MeDIP-seq, ChIP-seq, RNA-seq, microarray, PCR, and multicolor Flow Cytometry staining. DNA samples from the AREDS study, held under the DCR/NEI Repository protocol (07-EI-0168), will also be used for analysis. If necessary, the gene product or blood sample will be characterized biochemically.

Outcome Measures:

Immunophenotyping, gene expression and epigenetic changes will be reported using Statistical analysis performed using the t test or ANOVA and post-hoc testing with Fisher s least significant difference test. Unless otherwise noted, results are presented as the mean SEM. Biochemical, metabolic, and physiological effects will be individualized to the specific assay

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants with the following will be recruited:

* Individuals or family members of individuals with immune mediated retinal disorders, including uveitis, age related macular degeneration, and diabetic retinopathy.
* Adults must be capable of providing their own consent.
* All participants must be able to cooperate with study examination and phlebotomy.
* Children must be older than 4 years of age.

EXCLUSION CRITERIA:

* Individuals with diseases, infections, or trauma that mimic immune medicated retinal disorders.
* Children requiring sedation for study procedures.

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 609 (Actual)
Dates: Start 2008-03-27; Study Completion 2018-12-04

CONTACTS AND LOCATIONS:
Overall Officials: Hatice N Sen, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Becker KG, Simon RM, Bailey-Wilson JE, Freidlin B, Biddison WE, McFarland HF, Trent JM. Clustering of non-major histocompatibility complex susceptibility candidate loci in human autoimmune diseases. Proc Natl Acad Sci U S A. 1998 Aug 18;95(17):9979-84. doi: 10.1073/pnas.95.17.9979. PMID 9707586
- [Background] Richardson B. Primer: epigenetics of autoimmunity. Nat Clin Pract Rheumatol. 2007 Sep;3(9):521-7. doi: 10.1038/ncprheum0573. PMID 17762851
- [Background] Carrel L, Willard HF. X-inactivation profile reveals extensive variability in X-linked gene expression in females. Nature. 2005 Mar 17;434(7031):400-4. doi: 10.1038/nature03479. PMID 15772666